CLINICAL TRIAL: NCT02018120
Title: Comparison of Platelet Rich Fibrin and Connective Tissue Graft in Treatment of Multiple Gingival Recessions
Brief Title: Platelet Rich Fibrin in the Treatment of Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Asude Merve Polat, PhD, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-Dis-004
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Gingival Recession
Keywords: multiple gingival recession; platelet rich fibrin; connective tissue graft; microsurgery; periodontal diseases; gingival recession
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- connective tissue graft (Active Comparator): connective tissue graft harvested from palatum of subjects and placed under modified coronally advanced flap
  Interventions: Procedure: connective tissue graft
- Platelet rich fibrin (Experimental): Autogenous platelet rich fibrin was obtained from subjects own blood samples after centrifugation. Platelet rich fibrin membranes were placed under modified coronally advanced flaps.
  Interventions: Procedure: platelet rich fibrin

INTERVENTIONS:
Procedure: connective tissue graft
  Arms: connective tissue graft
Procedure: platelet rich fibrin
  Arms: Platelet rich fibrin

SUMMARY:
The aim of this randomized controlled clinical study is to evaluate and compare the effectiveness of platelet rich fibrin (PRF) and connective tissue grafts in the treatment of multiple gingival recessions.

DETAILED DESCRIPTION:
The aim of this randomized controlled clinical study is to evaluate and compare the effectiveness of platelet rich fibrin (PRF) and connective tissue grafts in the treatment of multiple gingival recessions.

Primary outcome variables were percentage of complete root coverage and mean root coverage percentages at 6 months follow up. The secondary outcome variables include keratinized tissue and gingival thickness gain.

Sample size has been estimated as 13 in each treatment arm. All recessions are treated with modified coronally advanced flap. On test sites PRF membrane and on control sites connective tissue grafts will be placed under modified coronally advanced flaps. Random allocation of the treatment sites to test and control groups were performed using a computer software designed for randomization.

Clinical parameters such as gingival index, plaque index, keratinized tissue width, gingival recession depth and width were measured at 1, 3 and 6 months. Probing pocket depth, clinical attachment level, gingival thickness and gingival recession area were measure at baseline and 6 months. All gingival recession-related parameters such as recession height, recession width and recession area and keratinized tissue width along with mean root coverage and complete root coverage were assessed on standardized clinical photographs using an image analysis software.

Clinical photographs were obtained at baseline and 1, 3 and 6 months after surgical intervention. 4 mm length wire was placed on gingiva to check reproducibility and to obtain standardized pictures.

Gingival tissue thickness were measured with an #15 endodontic reamer attached to rubber stopper inserted perpendicularly into the gingival tissue 2 mm below the gingival margin; thickness of the reamer will be measured with a digital caliper.

Mean root coverage percentage was calculated as percentage of covered root surface area at 6 months.

Follow up of subjects was 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Two or more adjacent teeth with at least 2 mm Miller Class I gingival recessions at non-molar teeth
* Identifiable CEJ on all teeth
* Age ≥ 18
* Presence of tooth vitality and absence of restorations and superficial caries in the treatment area
* No past surgical treatment history of affected area.
* Gingival thickness ≥ 0,8 mm for recession areas.
* Sufficient palatal donor tissue for connective tissue harvesting.

Exclusion Criteria:

* Smoking
* Pregnancy or lactation
* Systematic diseases that may affect outcomes of periodontal therapy
* Self-reported antibiotic medication within three months
* Occlusal trauma in treatment site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean root coverage percentage | 6 months
  mean area of root coverage achieved by surgical root coverage therapy.
complete root coverage percentage | 6 months
  percentage of gingival recession defects completely covered by flaps after 6 months

SECONDARY OUTCOMES:
keratinized tissue width | 6 months
  changes in keratinized tissue width at 6 months
gingival tissue thickness | 6 months
  changes from baseline in gingival tissue thickness at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gül Atilla, Professor, Study Director — Ege University School of Dentistry
Locations (1):
- Ege University School of Dentistry Department of Periodontology, Izmir, Bornova, Turkey (Türkiye)